CLINICAL TRIAL: NCT02411474
Title: Tear Cytokine Analysis as a Prediction or Diagnostic Marker in Ocular GvHD
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0008
Record Dates: First submitted 2015-03-05; First posted 2015-04-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Graft-versus-host Disease
Keywords: stem cell transplantation (SCT)
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — TEAR
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- With or without newly diagnosed chronic GVHD after SCT: The patients developed chronic GVHD after SCT/ The patients did not developed chronic GVHD after SCT

SUMMARY:
Investigate the profiles of tear cytokines in patients who underwent stem cell transplantation (SCT) and attempted to determine the applicability of tear cytokines in the diagnosis of chronic graft-versus-host disease (GVHD). Evaluate tear cytokines as biomarkers of chronic ocular GVHD severity.

ELIGIBILITY:
Inclusion Criteria:

* The patients patients aged 20-60 years who visited the clinic 3-12 months after SCT were included in the study.

Exclusion Criteria:

* The patients with histories of ocular surgery; ocular injury; and ocular diseases such as ocular infection, allergy, and autoimmune disease, as well as patients with long-term use of topical ocular medications except artificial tears.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male or non-pregnant female patients aged 20-60 years who visited the clinic 3-12 months after SCT were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
tear cytokine | 3-12 month after SCT
  comparison of tear cytokines (IL-2,4,10,17a, INF-r, TNF-a) concentrations in patients with or without newly diagnosed chronic GVHD after SCT using a multiplex immunobead assay
ocular surface status | 3-12 month after SCT
tear film break-up time | 3-12 month after SCT
conjunctival injection | 3-12 month after SCT
Schirmer's test I | 3-12 month after SCT
ocular surface disease index | 3-12 month after SCT

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Fraser CJ, Bhatia S, Ness K, Carter A, Francisco L, Arora M, Parker P, Forman S, Weisdorf D, Gurney JG, Baker KS. Impact of chronic graft-versus-host disease on the health status of hematopoietic cell transplantation survivors: a report from the Bone Marrow Transplant Survivor Study. Blood. 2006 Oct 15;108(8):2867-73. doi: 10.1182/blood-2006-02-003954. Epub 2006 Jun 20. PMID 16788100